CLINICAL TRIAL: NCT03796390
Title: Study Evaluating Safety and Efficacy of CAR-T Cells Targeting CD123 in Patients With Acute Myelocytic Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Collaborators: Hebei Yanda Ludaopei Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Daopei CD123CAR-T
Record Dates: First submitted 2019-01-04; First posted 2019-01-08 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Acute Myelocytic Leukemia
Keywords: AML，CD123
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD123 CAR-T cells (Experimental): Patients will be be treated with CD123 CAR-T cells
  Interventions: Biological: CD123 CAR-T cells

INTERVENTIONS:
Biological: CD123 CAR-T cells — Patients will be drawn 50-100 ml blood to obtain enough peripheral blood mononuclear cells (PBMC) for CAR-T manufacturing. The T cells will be purified from the PBMC, transduced with CAR lentiviral vector, expanded in vitro and then frozen for future administration. Chemotherapy will then be given. Following tumor burden reassessment, CD123 CAR-T cells will be infused.

SUMMARY:
This is an open, single-arm, phase I clinical study to evaluate efficacy and safety of chimeric antigen receptor T cell immunotherapy (CAR-T) targeting CD123 in the treatment of Acute Myelocytic Leukemia. A total of 15 patients are planned to be enrolled following up one year.

DETAILED DESCRIPTION:
Chimeric antigen receptor (CAR)-modified T cells targeted against CD19 have demonstrated unprecedented successes in treating patients with hematopoietic and lymphoid malignancies. Besides CD19, many other molecules such as CD22, CD30,BCMA,CD123, etc. may be potential in developing the corresponding CAR-T cells to treat patients whose tumors expressing those markers. In this study, investigators will evaluate the safety and efficacy of CAR-T targeting CD123 in patients with Acute Myelocytic Leukemia. The primary goal is safety assessment including cytokine storm response and any other adverse effects. In addition, disease status after treatment will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with acute myeloid leukemia who voluntarily signed informed consent and met the following criteria:

  1. Diagnosed as recurrent or refractory acute myeloid leukemia
  2. Tumor cells confirmed CD123 positive by Flow cytometry (FCM) or immunohistochemical detection, and CD123 positive rate >80%
  3. Age ≥ 2 years old, and <65 years old
  4. Estimated survival time is longer than 3 months from the date of signing the informed consent form
  5. KPS ≥ 80 points
  6. Important organs function need to meet the following conditions:

  1) EF>50%, and there is no obvious abnormality in ECG; 2) SpO2≥90%; 3)Cr≤2.5ULN; 4)ALT and AST≤4ULN, TBil≤50μmol/L 7. Subjects with a pregnancy plan must agree to take contraception before the enrollment study and after the study lasts for six months; if the subject is pregnant or suspects of pregnancy, the investigator should be notified immediately 8. Need to stop chemotherapy for at least 2 weeks before collecting the blood to manufacture CAR-T cells.

  9. For allogeneic hematopoietic stem cell transplantation subjects, it is necessary to stop the immunosuppressant against GVHD for at least 2 weeks before collecting autologous blood preparation, and if the donor is preparing blood, it is of no influence; 10. If the subject has a history of central nervous system (CNS) leukemia, the tumor cells in the cerebrospinal fluid need to be cleared and the white blood cell count <5 * 10^6 / L ,then can proceed lymphodepletion 11. Subjects who participate in other studies must withdraw other studies for 2 weeks before they can be enrolled.

Exclusion Criteria:

1. Combine other diseases not effectively controlled, including but not limited to persistent or poorly controlled infections, symptomatic congestive heart failure, unstable angina, arrhythmia, poorly controlled lung disease or mental illness
2. There are other active malignant tumors
3. Combined serious infection and can not be effectively controlled
4. Active hepatitis (HBV DNA or hepatitis C virus ribonucleic acid [HCVRNA] detection positive)
5. Human immunodeficiency virus (HIV) infection or syphilis infection
6. Have a history of severe allergies in biological products (including antibiotics)
7. One month after discontinuation of immunosuppressants, allogeneic hematopoietic stem cell transplantation patients still have acute graft versus host response (GvHD)
8. Female subjects are pregnant or lactating
9. Systemic administration of glucocorticoids within one week prior to CAR-T treatment
10. In the past, there was a prolonged QT interval or severe heart disease.
11. Active autoimmune diseases requiring systemic immunosuppressive therapy
12. The investigator believes that it may increase the risk of the subject or interfere with the study results.

Exit criteria：

1. The subjects request to withdraw from the study before CAR-T infusion
2. The subjects seriously violate the protocol
3. Before CAR-T infusion, the following indicators are still abnormal after treatment:

1) EF>50%, and there is no obvious abnormality in ECG 2) SpO2≥90% 3)Cr≤2.5ULN(the upper limit of normal ) 4) ALT and AST ≤ 4ULN, TBil ≤ 50μmol / L 4.Not enough T cells for manufacture standard CAR-T cells 5. Other serious adverse events occurred

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-12-26 (Actual); Primary Completion 2020-11-06 (Estimated); Study Completion 2021-06-06 (Estimated)

PRIMARY OUTCOMES:
Tumor load | Up to 12 months
  Tumor load will be quantified with radiology, bone marrow and/or blood samples dependent on diagnosis.

SECONDARY OUTCOMES:
CAR-T cell persistence | Up to 12 months
  CAR-T cell persistence will be quantified with flow cytometry and qPCR； Percentage of CART cells in BM and copies of car per ug DNA

CONTACTS AND LOCATIONS:
Overall Officials: Peihua Lu, PhD&MD, Study Chair — Hebei Yanda Ludaopei Hospital
Locations (1):
- Hebei Yanda Ludaopei Hospital, Langfang, Hebei, China